CLINICAL TRIAL: NCT02519777
Title: A Randomized, Double-Blinded, Placebo-Controlled Trial Comparing Antiretroviral Intensification With Maraviroc and Dolutegravir With No Intensification or Intensification With Dolutegravir Alone for the Treatment of Cognitive Impairment in HIV
Brief Title: Integrase and Maraviroc Intensification in Neurocognitive Dysfunction (InMIND)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A5324; 11909 (Registry Identifier: DAIDS-ES); NCT02406196 (obsolete NCT alias)
Record Dates: First submitted 2015-08-06; First posted 2015-08-11 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: HIV Infections
Keywords: HIV-Associated Neurocognitive Disorder
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc; dolutegravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Placebo MVC and placebo DTG (Placebo Comparator): In addition to their existing ART regimens, participants in Arm A received placebo for MVC and placebo for DTG.
  Interventions: Drug: Placebo for maraviroc (MVC); Drug: Placebo for dolutegravir (DTG)
- Arm B: DTG and placebo MVC (Experimental): In addition to their existing ART regimens, participants in Arm B received DTG and placebo for MVC.
  Interventions: Drug: Placebo for maraviroc (MVC); Drug: Dolutegravir (DTG)
- Arm C: MVC and DTG (Experimental): In addition to their existing ART regimens, participants in Arm C received MVC and DTG
  Interventions: Drug: Dolutegravir (DTG); Drug: Maraviroc (MVC)

INTERVENTIONS:
Drug: Placebo for maraviroc (MVC) — Administered orally as one 150 mg tablet BID OR two 300 mg tablet BID OR one 300 mg tablet BID depending upon background ARV regimen
  Arms: Arm A: Placebo MVC and placebo DTG; Arm B: DTG and placebo MVC
Drug: Placebo for dolutegravir (DTG) — Administered orally as one 50 mg tablet BID OR one 50 mg tablet QD depending upon background ARV regimen
  Arms: Arm A: Placebo MVC and placebo DTG
Drug: Dolutegravir (DTG) — Administered orally as one 50 mg tablet BID OR one 50 mg tablet QD depending upon background ARV regimen
  Arms: Arm B: DTG and placebo MVC; Arm C: MVC and DTG
Drug: Maraviroc (MVC) — Administered orally as one 150 mg tablet BID OR two 300 mg tablet BID OR one 300 mg tablet BID depending upon background ARV regimen
  Arms: Arm C: MVC and DTG

SUMMARY:
People infected with HIV often have cognitive dysfunction even if they are on antiretroviral therapy (ART) and have undetectable viral loads. The study evaluated if the addition of maraviroc (MVC) and dolutegravir (DTG) (which are two antiretroviral [ARV] medications) to participants' existing ART regimens improved participants' neurocognitive performance.

DETAILED DESCRIPTION:
HIV-infected people often have cognitive dysfunction (HIV-associated neurocognitive disorder, or HAND), which includes asymptomatic neurocognitive impairment (ANI), mild neurocognitive disorder (MND), and HIV-associated dementia (HAD), even if they are on ART and have undetectable viral loads. In this study, researchers evaluated the effectiveness of adding MVC and DTG to the current ART regimen of HIV-infected people with undetectable (<50 copies/mL) plasma HIV-1 RNA who had neurocognitive impairment and who had been on stable ART for at least 6 months prior to study entry. The purpose of this study was to evaluate if the addition of MVC and DTG to participants' existing ART regimens improved participants' neurocognitive performance.

Participants were randomly assigned to one of three arms. All participants remained on their existing ART regimens; they took their assigned study drugs in addition to their ART regimen. Study visits occurred at entry and Weeks 2, 4, 12, 24, 48, 72, and 96. Visits may have included physical examinations, blood collection, neurocognitive testing, pregnancy testing, and questionnaires. Some participants may have had an optional lumbar puncture procedure at study entry and Week 48. Participants returned for refills of study drugs on Weeks 36, 60, and 84.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by:

  * a licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen or plasma HIV-1 RNA viral load. NOTE: The term "licensed" refers to a United States Food and Drug Administration (FDA)-approved kit, which is required for all IND studies, or for sites located in countries other than the United States, a kit that has been certified or licensed by an oversight body within that country and validated internally. Non-US sites are encouraged to use US FDA-approved methods for IND studies. WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (eg, indirect versus competitive), or a Western blot or a plasma HIV-1 RNA. OR
  * Documentation of HIV diagnosis in the medical record by a healthcare provider.
* On current ART for at least 6 months prior to study entry with no interruption in treatment of greater than or equal to 7 consecutive days. Note: The following ART changes are allowed:

  * Tenofovir disoproxil fumarate (TDF) to tenofovir alafenamide fumarate (TAF)/TAF-containing fixed-dose combination regimens
  * Ritonavir (RTV) to cobicistat (COBI)/COBI-containing fixed-dose combination regimens
* No plans to change ART while on study. Note: The following planned ART changes are allowed:

  * TDF to TAF/TAF-containing fixed-dose combination regimens
  * RTV to COBI/COBI-containing fixed-dose combination regimens
* HIV-1 plasma RNA less than 50 copies/mL obtained within 90 days prior to study entry by any FDA-approved assay at any United States laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent, or at any network-approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance programs.
* No more than one HIV-1 plasma RNA greater than or equal to 50 and less than 200 copies/mL (only one "blip") in the past 6 months with a subsequent HIV-1 plasma RNA less than 50 copies/mL. NOTE: There should be no plasma HIV-1 RNA greater than 200 copies/mL within the 6 months prior to study entry.
* HAND diagnosis (ANI, MND, or HAD) within 60 days prior to study entry. HAND is defined as at least mild impairment on neurocognitive testing (more than one standard deviation below appropriate normative data in two domains of functioning) and no severely confounding factors.
* Screening laboratory values obtained within 60 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent, or at any network-approved non-US laboratory that operates in accordance with GCLP and participates in appropriate external quality assurance programs:

  * Absolute neutrophil count (ANC) greater than or equal to 500/mm^3
  * Hemoglobin greater than or equal to 7.5 g/dL
  * Platelet count greater than or equal to 40,000/mm^3
  * Creatinine less than or equal to 2.0 x upper limit of normal (ULN)
  * Aspartate transaminase (AST) less than or equal to 5 x ULN
  * Alanine transaminase (ALT) less than 3 x ULN
  * Alkaline phosphatase less than or equal to 5 x ULN
  * Total bilirubin less than 1.5 x ULN. NOTE: If the potential participant is taking an indinavir (IDV)- or atazanavir (ATV)-containing regimen at the time of screening, total bilirubin less than or equal to 5 x ULN is acceptable.
  * Creatinine clearance (CrCl) greater than or equal to 60 mL/min, either measured or estimated by Cockcroft-Gault equation. NOTE: A calculator for estimating the CrCl can be found at www.fstrf.org/ACTG/ccc.html
* Females of reproductive potential (women who have not been post-menopausal for at least 24 consecutive months, ie, who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, hysterectomy or bilateral salpingectomy or bilateral oophorectomy or tubal ligation) must have a negative serum or urine pregnancy test by any US clinic or laboratory that has a CLIA certification or its equivalent, or is using a point of care (POC) / CLIA-waived test, or at any network-approved non-US laboratory or clinic that operates in accordance with GCLP and participates in appropriate external quality assurance programs within 48 hours prior to study entry
* Females of reproductive potential must agree not to participate in the conception process (ie, active attempt to become pregnant, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, must use at least one reliable form of contraception. Female participants must use contraceptives while receiving study treatment and for 6 weeks after stopping study treatment. More information on this criterion is available in the protocol.
* Ability and willingness of participant to complete the neuropsychological tests
* Ability and willingness of participant or a legally authorized representative (see protocol for more information) to provide informed consent
* Ability and willingness to take oral study medications

Exclusion Criteria:

* Current or past medical condition(s) that in the opinion of the investigator prevents attribution of the cause of cognitive impairment to HIV. For example:

  * Major depressive disorder with psychotic features
  * Traumatic Brain Injury (TBI) with a clear impact on activities of daily living
  * Developmental delay, intellectual deficit, and/or severe educational disability resulting in some dependence for activities of daily living
  * Ongoing substance use disorder with significant impact on activities of daily living. Difficult or impossible to determine whether cognitive or functional decline is due to substance use or HIV, or both
  * Evidence of intoxication or withdrawal during the screening evaluation
  * Central nervous system (CNS) infections or opportunistic conditions: brain abscess (bacterial, mycobacterial, fungal or Toxoplasma), meningitis with persistent neurologic impairment, primary CNS lymphoma, progressive multifocal leukoencephalopathy (PML), or another structural brain lesion with neurological sequelae
  * Other CNS conditions: non-opportunistic primary or metastatic brain tumors, uncontrolled seizure disorder, progressive multiple sclerosis, stroke with neurological sequelae, or dementia due to causes other than HIV (eg, Alzheimer's disease)
  * Constitutional illness (eg, persistent unexplained fever, diarrhea, significant weight loss, disabling weakness) within 30 days of screening
  * Known untreated B12 deficiency or malnutrition (body mass index [BMI] less than 18) at screening
* Evidence of current hepatitis C virus infection (HCV) (ie, HCV antibody [Ab] positive within 90 days prior to study entry unless also shown to be plasma HCV RNA negative within the same time period)
* Unstable and advanced liver disease (as defined by the presence of at least one of the following: ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice)
* Prior or current use of any CCR5 antagonist (such as MVC and cenicriviroc [CVC]) and integrase inhibitor (such as RAL, DTG, and elvitegravir [EVG])
* Current use of any medication, including antiretrovirals, prohibited in the study (refer to the A5324 protocol-specific web page [PSWP] for the prohibited medications)
* Breastfeeding
* Presence of an AIDS-defining opportunistic infection within 6 months prior to entry. Note: Refer to the A5324 Manual of Operations (MOPS) for the list of AIDS-defining opportunistic infections.
* Active syphilis or treatment for syphilis within 90 days prior to study entry. NOTE: Active syphilis is defined as four-fold increase in serum rapid plasma reagin (RPR) or venereal disease research laboratory (VDRL) tests in an individual with past syphilis, or newly reactive serum RPR or VDRL with a reactive confirmatory test (enzyme immunoassays [EIA] or chemiluminescent assay [CIA], T. pallidum particle agglutination [TP-PA], or fluorescent treponemal antibody absorbed [FTA-ABS]).
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Robertson, PhD, Study Chair — University of North Carolina
Locations (30):
- United States (23):
  - UCLA CARE Center CRS, Los Angeles, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Harbor-UCLA CRS, Torrance, California
  - Whitman-Walker Health CRS, Washington D.C., District of Columbia
  - Northwestern University CRS, Chicago, Illinois
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS, Greensboro, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Case Clinical Research Site, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Trinity Health and Wellness Center CRS, Dallas, Texas
  - Houston AIDS Research Team CRS, Houston, Texas
  - University of Washington AIDS CRS, Seattle, Washington
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro, Brazil
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico
- South Africa (3):
  - Wits Helen Joseph Hospital CRS (Wits HJH CRS), Johannesburg, Gauteng
  - Durban International Clinical Research Site CRS, Durban, KwaZulu-Natal
  - Famcru Crs, Tygerberg, Western Cape
- Thailand (2):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Bangkok
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai

REFERENCES:
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 30 Clinical Research Sites (CRSs) in the United States, Thailand, Brazil, and South Africa between April 2016 and November 2018.
Period: Overall Study
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Started | 63 | 67 | 61
Completed | 57 | 59 | 57
Not Completed | 6 | 8 | 4
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 4 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Severe Debilitation | 1 | 1 | 1
Not completed — Not able to get to clinic | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All participants were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG | Total
Number analyzed (Participants) | 63 | 67 | 61 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (7) | 52 (9) | 52 (8) | 52 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 23 | 18 | 56
  Male | 48 | 44 | 43 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 17 | 10 | 42
  Not Hispanic or Latino | 48 | 50 | 51 | 149
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 5 | 6 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 30 | 30 | 37 | 97
  White | 23 | 29 | 16 | 68
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 3 | 1 | 1 | 5
Normalized Neurocognitive Test Scores [Mean (Standard Deviation); unit: total neurocognitive z-score] — The normalized neurocognitive test score (total z-score) was defined as the average of z-scores on a series of tests. Domestic participants took 14 Tests, while International Participants took 11 tests. Z-scores were calculated using a demographically appropriate norming process. Higher total z-scores correspond with better neurocognitive performance. Change was calculated as the total z-score at Week 48 minus the total z-score at Baseline.
  total neurocognitive z-score | -0.96 (0.79) | -0.97 (0.70) | -1.09 (0.70) | -1.00 (0.73)
CD4 Cell Count [Mean (Standard Deviation); unit: cells/mm^3] | 681 (294) | 703 (278) | 726 (331) | 703 (300)
CD8 Cell Count [Mean (Standard Deviation); unit: cells/mm^3] | 789 (334) | 809 (393) | 816 (393) | 805 (373)
HIV RNA [Count of Participants; unit: Participants]
  <50 copies/mL | 62 | 64 | 58 | 184
  ≥50 copies/mL | 1 | 3 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Normalized Composite Neurocognitive Test Score at Week 48 From Baseline
Description: The normalized composite neurocognitive test score (total z-score) was defined as the average of the z-scores from the following tests:
  Domestic (US-based) and International Participants:
  * Grooved pegboard dominant
  * Grooved pegboard non-dominant
  * Hopkins Verbal Learning Test (HVLT-R) Learning trials
  * HVLT-R Delayed recall
  * HVLT-R Delayed recognition
  * Semantic verbal fluency
  Domestic only:
  * Stroop color naming
  * Stroop word reading
  * Stroop interference trial
  * Letter fluency
  * Trail Making A
  * Trail Making B
  * WAIS-III Symbol search
  * Digit Symbol
  International only:
  * Timed Gait
  * Finger Tapping Dominant
  * Finger Tapping Non-dominant
  * Color Trail 1
  Z-scores were calculated using a demographically appropriate norming process. Higher z-scores correspond with better neurocognitive performance. Change was calculated as the total z-score at Week 48 minus the total z-score at Baseline.
Time Frame: Measured at Baseline and Week 48
Population: All participants who started study treatment were included in the analysis. Analysis performed under intention to treat (ITT) principle, all eligible randomized participants were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: total neurocognitive z-score
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 63 | 67 | 60
total neurocognitive z-score | 0.20 [0.02 to 0.37] | 0.26 [0.11 to 0.40] | 0.31 [0.16 to 0.46]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in normalized composite neurocognitive test scores at Week 48 from baseline; Test type: Superiority; p = 0.60, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in normalized composite neurocognitive test scores at Week 48 from baseline; Test type: Superiority; p = 0.33, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in normalized composite neurocognitive test scores at Week 48 from baseline; Test type: Superiority; p = 0.61, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Treatment Related Adverse Events (AEs)
Description: Treatment Related Adverse Events were determined by the study sites indicating a relationship between an adverse event and the study treatment.
Time Frame: Measured from treatment initiation through Week 96
Population: All participants who were randomized were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 63 | 67 | 61
Participants | 3 | 5 | 7

3. Secondary Outcome: Change in Normalized Composite Neurocognitive Test Score at Weeks 24, 72, and 96 From Baseline
Description: The normalized composite neurocognitive test score (total z-score) was defined as the average of the z-scores from the following tests:
  Domestic and International Participants:
  * Grooved pegboard dominant
  * Grooved pegboard non-dominant
  * HVLT-R Learning trials
  * HVLT-R Delayed recall
  * HVLT-R Delayed recognition
  * Semantic verbal fluency
  Domestic only:
  * Stroop color naming
  * Stroop word reading
  * Stroop interference trial
  * Letter fluency
  * Trail Making A
  * Trail Making B
  * WAIS-III Symbol search
  * Digit Symbol
  International only:
  * Timed Gait
  * Finger Tapping Dominant
  * Finger Tapping Non-dominant
  * Color Trail 1
  * Color Trail 2
  Z-scores were calculated using a demographically appropriate norming process. Higher z-scores correspond with better neurocognitive performance. Change was calculated as the total z-score at the given time point minus the total z-score at Baseline.
Time Frame: Measured at Baseline and Weeks 24, 72, and 96
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: total neurocognitive z-score
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 63 | 67 | 60
total neurocognitive z-score
  Change of Normalized Composite Neurocognitive Test Score (Week 24) | 0.14 [-0.02 to 0.30] | 0.18 [0.08 to 0.28] | 0.20 [0.07 to 0.33]
  Change of Normalized Composite Neurocognitive Test Score (Week 72) | 0.29 [0.12 to 0.45] | 0.32 [0.19 to 0.46] | 0.37 [0.23 to 0.50]
  Change of Normalized Composite Neurocognitive Test Score (Week 96) | 0.37 [0.19 to 0.55] | 0.34 [0.21 to 0.47] | 0.38 [0.23 to 0.52]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in normalized composite neurocognitive test scores at Week 24 from baseline; Test type: Superiority; p = 0.61, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in normalized composite neurocognitive test scores at Week 72 from baseline; Test type: Superiority; p = 0.72, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in normalized composite neurocognitive test scores at Week 96 from baseline; Test type: Superiority; p = 0.79, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in normalized composite neurocognitive test scores at Week 24 from baseline; Test type: Superiority; p = 0.55, t-test, 2 sided
Statistical Analysis 5: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in normalized composite neurocognitive test scores at Week 72 from baseline; Test type: Superiority; p = 0.47, t-test, 2 sided
Statistical Analysis 6: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in normalized composite neurocognitive test scores at Week 96 from baseline; Test type: Superiority; p = 0.95, t-test, 2 sided
Statistical Analysis 7: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in normalized composite neurocognitive test scores at Week 24 from baseline; Test type: Superiority; p = 0.85, t-test, 2 sided
Statistical Analysis 8: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in normalized composite neurocognitive test scores at Week 72 from baseline; Test type: Superiority; p = 0.67, t-test, 2 sided
Statistical Analysis 9: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in normalized composite neurocognitive test scores at Week 96 from baseline; Test type: Superiority; p = 0.70, t-test, 2 sided

4. Secondary Outcome: Change in Functional Status Scores
Description: Functional status scores were calculated based on the instrumental activities of daily living (IADLs) forms. IADL scores were calculated as the sum of the eight IADL tasks where the task scores were equal to 1 if a participant did not need assistance with the task and equal to 0 if a participant needed some level of help with the task. The maximum possible functional status score was 8, while the minimum possible functional status score was 0, with higher functional status scores indicating a higher level of functionality.
Time Frame: Measured at Baseline and Weeks 24, 48, 72, and 96
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 63 | 67 | 60
units on a scale
  Change from Baseline in IADL Score (Week 24) | 0.29 [-0.04 to 0.61] | 0.43 [0.07 to 0.80] | 0.15 [-0.19 to 0.49]
  Change from Baseline in IADL Score (Week 48) | 0.38 [0.12 to 0.64] | 0.45 [0.11 to 0.79] | 0.10 [-0.16 to 0.36]
  Change from Baseline in IADL Score (Week 72) | 0.40 [0.09 to 0.70] | 0.30 [-0.07 to 0.67] | 0.13 [-0.12 to 0.39]
  Change from Baseline in IADL Score (Week 96) | 0.16 [-0.21 to 0.53] | 0.28 [-0.08 to 0.64] | 0.20 [-0.13 to 0.53]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in functional status scores at Week 24 from baseline; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in functional status scores at Week 48 from baseline; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in functional status scores at Week 72 from baseline; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in functional status scores at Week 96 from baseline; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in functional status scores at Week 24 from baseline; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in functional status scores at Week 48 from baseline; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in functional status scores at Week 72 from baseline; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in functional status scores at Week 96 from baseline; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in functional status scores at Week 24 from baseline; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in functional status scores at Week 48 from baseline; Test type: Superiority; p = 0.80, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in functional status scores at Week 72 from baseline; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in functional status scores at Week 96 from baseline; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA Greater Than or Equal to 50 Copies/mL
Description: The number of participants with Plasma HIV-1 RNA greater than or equal to 50 copies/mL was assessed at each given time point.
Time Frame: Measured at Weeks 24, 48, and 96
Population: The analysis included all participants who started study treatment and had Plasma HIV-1 RNA measured at the scheduled study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 62 | 66 | 60
Participants
  HIV RNA (Week 24) | 3 | 1 | 1
  HIV RNA (Week 48): number analyzed (Participants) | 58 | 63 | 59
  HIV RNA (Week 48) | 3 | 0 | 1
  HIV RNA (Week 96): number analyzed (Participants) | 56 | 60 | 55
  HIV RNA (Week 96) | 1 | 6 | 2
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in number of participants with HIV-1 RNA ≥ 50 copies/mL at Week 24; Test type: Superiority; Difference in Percentage of Participants = 3.32, 95% CI 2-sided [-2.78 to 9.42]
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in number of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48; Test type: Superiority; Difference in Percentage of Participants = 5.17, 95% CI 2-sided [-0.53 to 10.87]
Statistical Analysis 3: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in number of participants with HIV-1 RNA ≥ 50 copies/mL at Week 96; Test type: Superiority; Difference in Percentage of Participants = -8.21, 95% CI 2-sided [-16.56 to 0.13]
Statistical Analysis 4: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in number of participants with HIV-1 RNA ≥ 50 copies/mL at Week 24; Test type: Superiority; Difference in Percentage of Participants = 3.17, 95% CI 2-sided [-3.07 to 9.42]
Statistical Analysis 5: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in number of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48; Test type: Superiority; Difference in Percentage of Participants = 3.48, 95% CI 2-sided [-3.11 to 10.06]
Statistical Analysis 6: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in number of participants with HIV-1 RNA ≥ 50 copies/mL at Week 96; Test type: Superiority; Difference in Percentage of Participants = -1.85, 95% CI 2-sided [-7.89 to 4.19]
Statistical Analysis 7: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in number of participants with HIV-1 RNA ≥ 50 copies/mL at Week 24; Test type: Superiority; Difference in Percentage of Participants = -0.15, 95% CI 2-sided [-4.53 to 4.23]
Statistical Analysis 8: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in number of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48; Test type: Superiority; Difference in Percentage of Participants = -1.69, 95% CI 2-sided [-4.99 to 1.60]
Statistical Analysis 9: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in number of participants with HIV-1 RNA ≥ 50 copies/mL at Week 96; Test type: Superiority; Difference in Percentage of Participants = 6.36, 95% CI 2-sided [-2.70 to 15.42]

6. Secondary Outcome: CD4+ T-cell Counts
Description: CD4+ T-cell counts were recorded at the given time point
Time Frame: Measured at Weeks 24, 48, and 96
Population: The analysis included all participants who started study treatment and had CD4+ T-cell counts measured at the scheduled study visits.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 63 | 67 | 60
cells/mm^3
  CD4 Count (Week 24): number analyzed (Participants) | 62 | 66 | 60
  CD4 Count (Week 24) | 660 [585 to 735] | 669 [610 to 727] | 773 [676 to 869]
  CD4 Count (Week 48): number analyzed (Participants) | 58 | 63 | 59
  CD4 Count (Week 48) | 638 [565 to 711] | 691 [628 to 754] | 758 [669 to 846]
  CD4 Count (Week 96): number analyzed (Participants) | 57 | 60 | 56
  CD4 Count (Week 96) | 674 [597 to 750] | 720 [648 to 793] | 788 [696 to 881]

7. Secondary Outcome: Change in CD4+ T-cell Count
Description: Changes in CD4+ T-cell count were calculated as the CD4+ T-cell count at a given time point minus the CD4+ T-cell count at Baseline.
Time Frame: Measured at Baseline and Weeks 24, 48, and 96
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 63 | 67 | 60
cells/mm^3
  Change from Baseline in CD4 Count (Week 24): number analyzed (Participants) | 62 | 66 | 60
  Change from Baseline in CD4 Count (Week 24) | -13 [-56 to 31] | -33 [-66 to -1] | 42 [-19 to 103]
  Change from Baseline in CD4 Count (Week 48): number analyzed (Participants) | 58 | 63 | 59
  Change from Baseline in CD4 Count (Week 48) | -43 [-82 to -5] | -19 [-61 to 23] | 21 [-28 to 69]
  Change from Baseline in CD4 Count (Week 96): number analyzed (Participants) | 57 | 60 | 56
  Change from Baseline in CD4 Count (Week 96) | -10 [-54 to 33] | 10 [-36 to 55] | 44 [-23 to 111]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in CD4+ T-cell count at Week 24 from baseline; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in CD4+ T-cell count at Week 48 from baseline; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in CD4+ T-cell count at Week 96 from baseline; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in CD4+ T-cell count at Week 24 from baseline; Test type: Superiority; p = 0.42, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in CD4+ T-cell count at Week 48 from baseline; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in CD4+ T-cell count at Week 96 from baseline; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in CD4+ T-cell count at Week 24 from baseline; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in CD4+ T-cell count at Week 48 from baseline; Test type: Superiority; p = 0.33, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in CD4+ T-cell count at Week 96 from baseline; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: CD8+ T-cell Counts
Description: CD8+ T-cell counts were recorded at the given time point
Time Frame: Measured at Weeks 24, 48, and 96
Population: The analysis included all participants who started study treatment and had CD8+ T-cell counts measured at the scheduled study visits.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 63 | 67 | 60
cells/mm^3
  CD8 Count (Week 24): number analyzed (Participants) | 62 | 66 | 60
  CD8 Count (Week 24) | 757 [684 to 830] | 752 [671 to 833] | 862 [748 to 976]
  CD8 Count (Week 48): number analyzed (Participants) | 58 | 63 | 59
  CD8 Count (Week 48) | 742 [655 to 828] | 731 [648 to 814] | 856 [759 to 954]
  CD8 Count (Week 96): number analyzed (Participants) | 57 | 60 | 56
  CD8 Count (Week 96) | 747 [664 to 830] | 773 [671 to 876] | 879 [776 to 983]

9. Secondary Outcome: Change in CD8+ T-cell Count
Description: Changes in CD8+ T-cell count were calculated as the CD8+ T-cell count at a given time point minus the CD8+ T-cell count at baseline.
Time Frame: Measured at Baseline and Weeks 24, 48, and 96
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 63 | 67 | 60
cells/mm^3
  Change from Baseline in CD8 Count (Week 24): number analyzed (Participants) | 62 | 66 | 60
  Change from Baseline in CD8 Count (Week 24) | -29 [-83 to 24] | -61 [-102 to -19] | 44 [-24 to 112]
  Change from Baseline in CD8 Count (Week 48): number analyzed (Participants) | 58 | 63 | 59
  Change from Baseline in CD8 Count (Week 48) | -45 [-111 to 22] | -82 [-133 to -31] | 35 [-32 to 103]
  Change from Baseline in CD8 Count (Week 96): number analyzed (Participants) | 57 | 60 | 56
  Change from Baseline in CD8 Count (Week 96) | -43 [-97 to 12] | -33 [-87 to 21] | 44 [-31 to 118]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in CD8+ T-cell count at Week 24 from baseline; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in CD8+ T-cell count at Week 48 from baseline; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in CD8+ T-cell count at Week 96 from baseline; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in CD8+ T-cell count at Week 24 from baseline; Test type: Superiority; p = 0.27, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in CD8+ T-cell count at Week 48 from baseline; Test type: Superiority; p = 0.23, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in CD8+ T-cell count at Week 96 from baseline; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in CD8+ T-cell count at Week 24 from baseline; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in CD8+ T-cell count at Week 48 from baseline; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in CD8+ T-cell count at Week 96 from baseline; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in Log10 sCD14 in Plasma at Week 48 From Baseline
Description: Changes in Log10 sCD14 in Plasma were calculated as the Log10 sCD14 in Plasma at Week 48 minus the Log10 sCD14 in Plasma at Baseline.
Time Frame: Measured at Baseline and Week 48
Population: The analysis population consisted of all participants who had plasma samples available at Baseline and Week 48.
Measure: Mean (95% Confidence Interval); unit: Log10 ng/mL
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 54 | 54 | 54
Log10 ng/mL | 0.04 [0.00 to 0.08] | 0.03 [-0.01 to 0.07] | 0.01 [-0.03 to 0.04]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in Log10 sCD14 in plasma at Week 48 from baseline; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in Log10 sCD14 in plasma at Week 48 from baseline; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in Log10 sCD14 in plasma at Week 48 from baseline; Test type: Superiority; p = 0.96, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in Log10 MIP-1 Beta in Plasma at Week 48 From Baseline
Description: Changes in Log10 MIP-1 Beta in Plasma were calculated as the Log10 MIP-1 Beta in Plasma at Week 48 minus the Log10 MIP-1 Beta in Plasma at Baseline. Results below the lower limit of quantification were set to the lower limit value of 11.
Time Frame: Measured at Baseline and Week 48
Population: The analysis population consisted of all participants who had plasma samples available at Baseline and Week 48
Measure: Mean (95% Confidence Interval); unit: Log10 pg/mL
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 54 | 54 | 54
Log10 pg/mL | 0.05 [-0.04 to 0.14] | -0.02 [-0.10 to 0.06] | 0.30 [0.22 to 0.37]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in Log10 MIP-1 Beta in plasma at Week 48 from baseline; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in Log10 MIP-1 Beta in plasma at Week 48 from baseline; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in Log10 MIP-1 Beta in plasma at Week 48 from baseline; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change in Log10 sTNFr-II in Plasma at Week 48 From Baseline
Description: Changes in Log10 sTNFr-II in Plasma were calculated as the Log10 sTNFr-II in Plasma at Week 48 minus the Log10 sTNFr-II in Plasma at Baseline.
Time Frame: Measured at Baseline and Week 48
Population: The analysis population consisted of all participants who had plasma samples available at Baseline and Week 48
Measure: Mean (95% Confidence Interval); unit: Log10 pg/mL
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 54 | 54 | 54
Log10 pg/mL | 0.02 [-0.02 to 0.05] | 0.01 [-0.02 to 0.04] | 0.00 [-0.04 to 0.03]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in Log10 sTNFr-II in plasma at Week 48 from baseline; Test type: Superiority; p = 0.91, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in Log10 sTNFr-II in plasma at Week 48 from baseline; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in Log10 sTNFr-II in plasma at Week 48 from baseline; Test type: Superiority; p = 0.94, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Change in Log10 VCAM in Plasma at Week 48 From Baseline
Description: Changes in Log10 VCAM in Plasma were calculated as the Log10 VCAM in Plasma at Week 48 minus the Log10 VCAM in Plasma at Baseline.
Time Frame: Measured at Baseline and Week 48
Population: The analysis population consisted of all participants who had plasma samples available at Baseline and Week 48
Measure: Mean (95% Confidence Interval); unit: Log10 pg/mL
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 54 | 54 | 54
Log10 pg/mL | 0.01 [-0.02 to 0.05] | 0.00 [-0.02 to 0.03] | 0.00 [-0.03 to 0.02]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in Log10 VCAM in plasma at Week 48 from baseline; Test type: Superiority; p = 0.70, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in Log10 VCAM in plasma at Week 48 from baseline; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in Log10 VCAM in plasma at Week 48 from baseline; Test type: Superiority; p = 0.85, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change in Log10 MIP-1 Beta in Cerebrospinal Fluid (CSF) at Week 48 From Baseline
Description: Changes in Log10 MIP-1 Beta in CSF were calculated as the Log10 MIP-1 Beta in CSF at Week 48 minus the Log10 MIP-1 Beta in CSF at Baseline.
Time Frame: Measured at Baseline and Week 48
Population: The analysis population consisted of all participants who had CSF samples available at Baseline and Week 48
Measure: Mean (95% Confidence Interval); unit: Log10 pg/mL
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 13 | 12 | 9
Log10 pg/mL | -0.24 [-0.71 to 0.23] | -0.32 [-0.77 to 0.14] | 0.17 [-0.42 to 0.76]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in Log10 MIP-1 Beta in CSF at Week 48 from baseline; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in Log10 MIP-1 Beta in CSF at Week 48 from baseline; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in Log10 MIP-1 Beta in CSF at Week 48 from baseline; Test type: Superiority; p = 0.20, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change in Log10 IP-10 in CSF at Week 48 From Baseline
Description: Changes in Log10 IP-10 in CSF were calculated as the Log10 IP-10 in CSF at Week 48 minus the Log10 IP-10 in CSF at Baseline.
Time Frame: Measured at Baseline and Week 48
Population: The analysis population consisted of all participants who had CSF samples available at Baseline and Week 48
Measure: Mean (95% Confidence Interval); unit: Log10 pg/mL
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 13 | 12 | 9
Log10 pg/mL | 0.02 [-0.06 to 0.09] | -0.11 [-0.33 to 0.10] | -0.36 [-0.99 to 0.26]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in Log10 IP-10 in CSF at Week 48 from baseline; Test type: Superiority; p = 0.59, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in Log10 IP-10 in CSF at Week 48 from baseline; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in Log10 IP-10 in CSF at Week 48 from baseline; Test type: Superiority; p = 0.80, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Change in Log10 Neopterin in CSF at Week 48 From Baseline
Description: Changes in Log10 Neopterin in CSF were calculated as the Log10 Neopterin in CSF at Week 48 minus the Log10 Neopterin in CSF at Baseline.
Time Frame: Measured at Baseline and Week 48
Population: The analysis population consisted of all participants who had CSF samples available at Baseline and Week 48
Measure: Mean (95% Confidence Interval); unit: Log10 nmol/L
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 13 | 12 | 9
Log10 nmol/L | 0.01 [-0.04 to 0.06] | -0.06 [-0.22 to 0.10] | -0.17 [-0.51 to 0.17]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in Log10 Neopterin in CSF at Week 48 from baseline; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in Log10 Neopterin in CSF at Week 48 from baseline; Test type: Superiority; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in Log10 Neopterin in CSF at Week 48 from baseline; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Change in Log10 NFL in CSF at Week 48 From Baseline
Description: Changes in Log10 NFL in CSF were calculated as the Log10 NFL in CSF at Week 48 minus the Log10 NFL in CSF at Baseline.
Time Frame: Measured at Baseline and Week 48
Population: The analysis population consisted of all participants who had CSF samples available at Baseline and Week 48
Measure: Mean (95% Confidence Interval); unit: Log10 pg/mL
Arm/Group | Arm A: Placebo MVC and Placebo DTG | Arm B: DTG and Placebo MVC | Arm C: MVC and DTG
Number analyzed (Participants) | 13 | 12 | 9
Log10 pg/mL | -0.02 [-0.08 to 0.05] | -0.05 [-0.12 to 0.02] | 0.00 [-0.14 to 0.14]
Statistical Analysis 1: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm B: DTG and Placebo MVC; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm B: DTG and placebo MVC in change in Log10 NFL in CSF at Week 48 from baseline; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm A: Placebo MVC and Placebo DTG vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm A: Placebo MVC and placebo DTG and Arm C: MVC and DTG in change in Log10 NFL in CSF at Week 48 from baseline; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm B: DTG and Placebo MVC vs Arm C: MVC and DTG; Under the null hypothesis, it was assumed there was no difference between Arm B: DTG and placebo MVC and Arm C: MVC and DTG in change in Log10 NFL in CSF at Week 48 from baseline; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)

18. Other Pre Specified Outcome: Changes in Cell-associated HIV-1 RNA/DNA/2-long Terminal Repeat Sequences (LTR) Circles and Single Copy Assay (SCA)
Description: This outcome measure was listed as secondary in the protocol but the intention was as an exploratory outcome due to lack of funding for testing.
Time Frame: Measured at Baseline and Week 48
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Changes in T Cell and Monocyte Activation
Description: as for outcome 18
Time Frame: Measured at Baseline and Week 48
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Changes in Residual Viremia
Description: as for outcome 18
Time Frame: Measured at Baseline and Week 48
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From treatment initiation to study completion at Week 96 or premature study discontinuation
Description: Post-entry, all new diagnoses, signs/symptoms and laboratory events of ≥ Grade 3 and all signs/symptoms and laboratory events that led to a change in treatment, regardless of grade, were collected. The DAIDS AE Grading Table (V2.1) and Expediated Adverse Events (EAE) Manual (V2.0) were used. All eligible participants who initiated study treatment are included.
Groups:
- Arm A (Placebo DTG/Placebo MVC): In addition to their existing ART regimens, participants in Arm A received placebo for MVC and placebo for DTG.
  Placebo for maraviroc (MVC): Administered orally as one 150 mg tablet BID OR two 300 mg tablet BID OR one 300 mg tablet BID depending upon background ARV regimen
  Placebo for dolutegravir (DTG): Administered orally as one 50 mg tablet BID OR one 50 mg tablet QD depending upon background ARV regimen
- Arm B (DTG/Placebo MVC): In addition to their existing ART regimens, participants in Arm B received DTG and placebo for MVC.
  Placebo for maraviroc (MVC): Administered orally as one 150 mg tablet BID OR two 300 mg tablet BID OR one 300 mg tablet BID depending upon background ARV regimen
  Dolutegravir (DTG): Administered orally as one 50 mg tablet BID OR one 50 mg tablet QD depending upon background ARV regimen
- Arm C (DTG/MVC): In addition to their existing ART regimens, participants in Arm C received MVC and DTG
  Dolutegravir (DTG): Administered orally as one 50 mg tablet BID OR one 50 mg tablet QD depending upon background ARV regimen
  Maraviroc (MVC): Administered orally as one 150 mg tablet BID OR two 300 mg tablet BID OR one 300 mg tablet BID depending upon background ARV regimen
Arm/Group | Arm A (Placebo DTG/Placebo MVC) | Arm B (DTG/Placebo MVC) | Arm C (DTG/MVC)
All-Cause Mortality (participants affected / at risk) | 1/63 | 0/67 | 0/60
Serious Adverse Events (participants affected / at risk) | 6/63 | 12/67 | 9/60
Other Adverse Events (participants affected / at risk) | 31/63 | 32/67 | 37/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Placebo DTG/Placebo MVC) (N=63) | Arm B (DTG/Placebo MVC) (N=67) | Arm C (DTG/MVC) (N=60)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Placebo DTG/Placebo MVC) (N=63) | Arm B (DTG/Placebo MVC) (N=67) | Arm C (DTG/MVC) (N=60)
Nausea (Gastrointestinal disorders) | 2 | 3 | 3
Chest pain (General disorders) | 0 | 0 | 4
Fatigue (General disorders) | 2 | 4 | 2
Pain (General disorders) | 0 | 1 | 3
Pyrexia (General disorders) | 3 | 4 | 3
Influenza (Infections and infestations) | 1 | 2 | 3
Alanine aminotransferase increased (Investigations) | 4 | 3 | 3
Aspartate aminotransferase increased (Investigations) | 5 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 6 | 6 | 5
Blood bicarbonate decreased (Investigations) | 1 | 2 | 3
Blood bilirubin increased (Investigations) | 3 | 7 | 5
Blood creatinine increased (Investigations) | 3 | 9 | 15
Blood glucose increased (Investigations) | 8 | 8 | 10
Blood phosphorus decreased (Investigations) | 6 | 4 | 2
Blood potassium decreased (Investigations) | 1 | 0 | 3
Blood sodium increased (Investigations) | 0 | 0 | 3
Creatinine renal clearance decreased (Investigations) | 2 | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (6):
  • Study Protocol and Informed Consent Form: Protocol V2.0 (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT02519777/Prot_ICF_000.pdf
  • Study Protocol: Protocol V2.0_Letter of Amendment 1 (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT02519777/Prot_001.pdf
  • Study Protocol: Protocol V2.0_Letter of Amendment 2 (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT02519777/Prot_002.pdf
  • Study Protocol: Protocol V2.0_Letter of Amendment 3 (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT02519777/Prot_003.pdf
  • Study Protocol: Protocol V2.0_Letter of Amendment 4 (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT02519777/Prot_004.pdf
  • Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT02519777/SAP_005.pdf